CLINICAL TRIAL: NCT02908750
Title: An Open-label, Non-randomised, Phase I Study to Assess the Effect of Single and Multiple Oral Doses of Osimertinib (TAGRISSO™) on the Pharmacokinetics of a P-glycoprotein Probe Drug (Fexofenadine) in Patients With Advanced EGFRm NSCLC That Have Progressed on a Prior EGFR-TKI Regimen
Brief Title: Study to Assess the Effect of Osimertinib (TAGRISSO™ ) on Blood Levels of Fexofenadine in Patients With EGFRm+ NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00036
Record Dates: First submitted 2016-08-23; First posted 2016-09-21 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: oncology; cancer; non small cell lung cancer; anticancer drug; lung neoplasms; pharmacokinetics; AZD9291; osimertinib; fexofenadine; TAGRISSO™; EGFR genes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms | interventions — Acetylcysteine; fexofenadine; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- osimertinib and fexofenadine (Experimental): Sequential treatments of fexofenadine alone followed by osimertinib + fexofenadine, followed by osimertinib alone, followed by osimertinib + fexofenadine
  Interventions: Drug: Fexofenadine tablet dosing; Drug: Osimertininb tablet dosing

INTERVENTIONS:
Drug: Fexofenadine tablet dosing — Fexofenadine (P-gp substrate) 120mg taken once daily on Days 1 in Treatment Period 1 and Day 1 and Day 39 in Treatment Period 2
  Other Names: Mucinex, Allegra, Select, Rugby
Drug: Osimertininb tablet dosing — Osimertininb 80 mg taken once daily on Day 1 and Days 4 to 41 in Treatment Period 2
  Other Names: TAGRISSO™

SUMMARY:
This is a Phase I, open-label, 2-part study in patients with a confirmed diagnosis of epidermal growth factor receptor (EGFR) mutation positive (EGFRm+) non-small cell lung cancer (NSCLC), who have progressed following prior therapy with an approved EGFR tyrosine kinase inhibitor (TKI) agent.

Part A will assess the effect of osimertinib on the pharmacokinetic (PK) parameters of fexofenadine, following single and multiple oral dosing of osimertinib in a fasted state.

Continuous Access will allow patients further access to osimertinib after the PK phase (Part A). All patients from Part A who completed treatment may continue to receive osimertinib 80 mg once daily until: they are no longer deriving clinical benefit; or any other reason

DETAILED DESCRIPTION:
This is a Phase I, open-label, non-randomised, two-part study in patients with EGFRm+ NSCLC who have progressed on an EGFR-TKI.

The PK phase will assess the effect of osimertinib on the PK parameters of fexofenadine following both single and multiple oral dosing of osimertinib. Continued access will provide patients with further access to osimertinib after the PK phase.

The study will be conducted at approximately 10 sites across Asia and Western Europe, with approximately 24 patients enrolled in order to achieve at least 18 evaluable patients. Additional patients may be dosed to ensure the minimum number of evaluable patients.

PK phase The PK phase is a non-randomised, open-label, 2-period design. Treatment Period 1 and Treatment Period 2 are separated by a 3 to 7 day washout period between doses. A study flow chart for the PK phase is presented in Figure 1. Patients will receive osimertinib 80 mg as a single dose on Day 1 of Treatment Period 2, then 80 mg once daily for 38 days (from Day 4 to Day 41 in Treatment Period 2). Patients will also receive a single oral dose of fexofenadine on Day 1 in Treatment Period 1, and on Days 1 and 39 in Treatment Period 2.

Continued access On completion of the PK phase (ie, following collection of the 72-hour fexofenadine sample on Day 42), patients may continue to take osimertinib tablets (80 mg once daily) as a single agent in continued access if they and the Investigator agree that this is appropriate. This will continue until the Investigator believes they are no longer deriving clinical benefit, or they stop taking osimertinib for any other reason. No clinical data will be collected during this phase other than sudden death of unknown reason, serious adverse events (SAEs) that may be related to osimertinib, outcomes of pregnancy and drug dispensing/accountability.

If a patient discontinues treatment during the PK phase, they will return to the clinic for follow-up assessments 30 days (±7 days) after their last dose of treatment in the PK phase. If the patient's last dose of osimertinib is in continued access, the patient should be contacted 30 days after their last dose of osimertinib to follow-up any existing SAEs, monitor for new SAEs that may be related to the IP, and record any sudden deaths of unknown cause.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 years
* Histological or cytological confirmation diagnosis of NSCLC
* Radiological documentation of disease progression while receiving previous continuous treatment with an EGFR-TKI.
* Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR-TKI sensitivity
* ECOG performance status 0 to 1, with no deterioration over the previous 2 weeks.
* Patients must have a life expectancy of 12 weeks or longer
* Females should be using adequate contraceptive measures and must have a negative serum pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child bearing potential.
* Male patients should be willing to use barrier contraception ie, condoms until 6 months after the last study drug is taken.
* For inclusion in optional genetic research, patients must provide separate informed consent.

Exclusion Criteria:

* Treatment with any of the following:

  * A 1st or 2nd generation EGFR-TKI within 8 days or approximately 5 half-lives, of the first dose of study treatment
  * Osimertinib in the present study [ie, dosing with osimertinib previously initiated in this study] or has previously received a 3rd generation EGFR-TKI [eg, CO 1686].
  * Any cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment.
  * Major surgery [excluding placement of vascular access] within 4 weeks of the first dose of study treatment.
  * Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment
  * Patients currently receiving [or unable to stop at least 3 weeks prior to first dose of osimertinib] medications or herbal supplements known to be potent inducers of CYP3A4 or inducers/inhibitors of P-gp.
* Spinal cord compression or brain metastases, unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval corrected for heart rate using Fridericia's correction factor [QTcF] greater than 470 msec, obtained from 3 ECGs.
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG [eg, complete left bundle branch block, third degree heart block, second degree heart block, PR interval greater than 250 msec]
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

  * Absolute neutrophil count [ANC] less than 1.5 × 109/L
  * Platelet count less than 100 × 109/L
  * Haemoglobin less than 90 g/L
  * ALT greater than 2.5 times ULN if no demonstrable liver metastases or greater than 5 times ULN in the presence of liver metastases
  * AST greater than 2.5 times ULN if no demonstrable liver metastases or greater than 5 times ULN in the presence of liver metastases
  * Total bilirubin greater than 1.5 times ULN if no liver metastases or greater than 3 times ULN in the presence of liver metastases
  * Creatinine greater than 1.5 times institutional ULN concurrent with creatinine clearance less than 50 mL/min [measured or calculated by Cockcroft-Gault formula]
* Patients unable to swallow orally administered medication or with gastrointestinal disorders or significant gastrointestinal resection likely to interfere with the absorption of the study drugs.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Fexofenadine Cmax (alone and in combination with osimertinib) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 24, 36, 48, 60, 72 on Day 1 in Period 1 and Day 1 and Day 39 in Period 2
  To characterize the pharmacokinetics of fexofenadine by assessment of maximum plasma fexofenadine concentration.
Fexofenadine AUC (alone and in combination with osimertinib) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 24, 36, 48, 60, 72 on Day 1 in Period 1 and Day 1 and Day 39 in Period 2.
  To characterize the pharmacokinetics of fexofenadine by assessment of area under the plasma concentration time curve from zero to infinity

SECONDARY OUTCOMES:
Fexofenadine tmax (alone and in combination with osimertinib) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 24, 36, 48, 60, 72 on Day 1 in Period 1 and Day 1 and Day 39 in Period 2
  To characterize the pharmacokinetics of fexofenadine by assessment of time to reach maximum plasma concentration
Fexofenadine AUC0-t (alone and in combination with osimertinib) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 24, 36, 48, 60, 72 on Day 1 in Period 1 and Day 1 and Day 39 in Period 2
  To characterize the pharmacokinetics of fexofenadine by assessment of area under plasma concentration-time curve from time zero to the last quantifiable time point
Fexofenadine CL/F (alone and in combination with osimertinib) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 24, 36, 48, 60, 72 on Day 1 in Period 1 and Day 1 and Day 39 in Period 2
  To characterize the pharmacokinetics of fexofenadine by assessment of apparent plasma clearance following oral administration
Fexofenadine Vz/F (alone and in combination with osimertinib) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 24, 36, 48, 60, 72 on Day 1 in Period 1 and Day 1 and Day 39 in Period 2
  To characterize the pharmacokinetics of fexofenadine by assessment of apparent volume of distribution
Fexofenadine λz (alone and in combination with osimertinib) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 24, 36, 48, 60, 72 on Day 1 in Period 1 and Day 1 and Day 39 in Period 2
  To characterize the pharmacokinetics of fexofenadine by assessment of terminal rate constant
Fexofenadine t½λz (alone and in combination with osimertinib) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 24, 36, 48, 60, 72 on Day 1 in Period 1 and Day 1 and Day 39 in Period 2
  To characterize the pharmacokinetics of fexofenadine by assessment of terminal half-life
Osimertinib and metabolites (AZ5104 and AZ7550) | Blood samples are collected pre-dose on D11, D18, D25, and D32
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of trough concentrations
Osimertinib and metabolites (AZ5104 and AZ7550) single dose: AUC0-72 | Blood samples are collected pre-dose, 1, 2, 3, 4, 5, 6, 8, 10 24, 36, 48, 60, 72 on Day 1 in Period 2
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of area under plasma concentration-time curve from time zero to 72 hours post-dose
Osimertinib and metabolites (AZ5104 and AZ7550) single dose: Cmax | Blood samples are collected pre-dose, 1, 2, 3, 4, 5, 6, 8, 10 24, 36, 48, 60, 72 on Day 1 in Period 2
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of maximum plasma drug concentration
Osimertinib and metabolites (AZ5104 and AZ7550) single dose: tmax | Blood samples are collected pre-dose, 1, 2, 3, 4, 5, 6, 8, 10 24, 36, 48, 60, 72 on Day 1 in Period 2
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of Time to reach maximum plasma concentration
Osimertinib and metabolites (AZ5104 and AZ7550) single dose: MRCmax | Blood samples are collected pre-dose, 1, 2, 3, 4, 5, 6, 8, 10 24, 36, 48, 60, 72 on Day 1 in Period 2
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of metabolite to parent ratio (AZ5104:osimertinib, AZ7550:osimertinib) maximum plasma drug concentration
Osimertinib and metabolites (AZ5104 and AZ7550) multiple dose: AUCtau | Blood samples are collected pre-dose, 1, 2, 3, 4, 5, 6, 8, 10 24 on Day 39 in Period 2
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of area under plasma concentration time curve during the dosing interval
Osimertinib and metabolites (AZ5104 and AZ7550) multiple dose Css,max | Blood samples are collected pre-dose, 1, 2, 3, 4, 5, 6, 8, 10 24 on Day 39 in Period 2
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of maximum plasma concentration at steady state
Osimertinib and metabolites (AZ5104 and AZ7550) multiple dose Css,min | Blood samples are collected pre-dose, 1, 2, 3, 4, 5, 6, 8, 10 24 on Day 39 in Period 2
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of minimum plasma concentration at steady state
Osimertinib and metabolites (AZ5104 and AZ7550) multiple dose: CLss/F (osimertinib only) | Blood samples are collected pre-dose, 1, 2, 3, 4, 5, 6, 8, 10 24 on Day 39 in Period 2
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of apparent plasma clearance following oral administration at steady state
Osimertinib and metabolites (AZ5104 and AZ7550) multiple doses: MRAUCtau | Blood samples are collected pre-dose, 1, 2, 3, 4, 5, 6, 8, 10 24 on Day 39 in Period 2
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of metabolite to parent ratio (AZ5104:osimertinib, AZ7550:osimertinib) area under plasma concentration time curve during the dosing interval
Osimertinib and metabolites (AZ5104 and AZ7550) multiple dose: MRCss,max | Blood samples are collected pre-dose, 1, 2, 3, 4, 5, 6, 8, 10 24 on Day 39 in Period 2
  To characterize the pharmacokinetics of osimertinib and metabolites (AZ5104 and AZ7550) by assessment of metabolite to parent ratio (AZ5104:osimertinib, AZ7550:osimertinib) maximum plasma concentration at steady state
Safety data collected using: Assessment of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Part A, approximately 11 weeks
Safety data collected using: Assessment of serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) (Version 4) | Part A and Continuous Access, approximately 24 months
Safety data collected using: vital signs (blood pressure, pulse, temperature, height, weight) | Part A, approximately 11 weeks
Safety data collected using: laboratory parameters (clinical chemistry, heamatology, urinalysis) | Part A, approximately 11 weeks
Safety data collected using: physical examination | Part A, approximately 11 weeks
Safety data collected using: standard 12-lead electrocardiograms (ECGS) | Part A, approximately 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano C Aller, M.D., Ph.D., Principal Investigator — Centro Integral Oncologico Clara Campal
Locations (5):
- Research Site, Rennes, France
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (2):
  - Research Site, Madrid
  - Research Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Calvo E, Lee JS, Kim SW, Moreno V, deCastro Carpeno J, Weilert D, Laus G, Mann H, Vishwanathan K. Modulation of Fexofenadine Pharmacokinetics by Osimertinib in Patients With Advanced EGFR-Mutated Non-Small Cell Lung Cancer. J Clin Pharmacol. 2019 Aug;59(8):1099-1109. doi: 10.1002/jcph.1403. Epub 2019 Mar 15. PMID 30875094
- See also: Redacted CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4200&filename=d5160c00036-csp-v1_Redacted.pdf